CLINICAL TRIAL: NCT02141945
Title: Metabiomics Neoplasia Clinical Research Study
Brief Title: Microbiome Test for the Detection of Colorectal Polyps and Cancer
Status: Completed | Type: Observational
Sponsor: Metabiomics Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: MB-01
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer
Keywords: Cancer; Colon Cancer; Colorectal Cancer; Neoplasm; Colorectal Neoplasm; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Colonic Diseases; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Colonic Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Colonic Diseases; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — gut microbiome samples from stool, rectal and colonic mucosa
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose if this study is to measure the sensitivity, specificity and accuracy of the Metabiomics Colon Polyp and Colorectal Cancer Assay for the non-invasive detection of colon polyps or colorectal cancer.

DETAILED DESCRIPTION:
The purpose of this study is to conduct clinical research to investigate the association of the gut microbiome with colonic neoplasia. In this study patients will supply samples of their gut microbiome prior to scheduled colonoscopy; the relative abundance of microbes from those samples will be used to predict the presence or absence of colon polyps or colorectal cancer. Microbiome based predictions from blinded samples will be compared with colonoscopy and pathology results to quantify the sensitivity, specificity and accuracy (reported as %) of the Metabiomics Colon Polyp and Colorectal Cancer Assay for colon polyps. The limited sample size is anticipated to be insufficient to quantify sensitivity to colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Age: 45-80 years,
* Patients undergoing polyp surveillance or screening colonoscopy who are ASA Class 1-3. No ASA Class 4 or 5 will be included.Footnote
* All ethnic and racial groups will be included,
* Able to comprehend, sign, and date the written informed consent form (ICF),
* Able to give informed consent in English.

Exclusion Criteria:

* History of Inflammatory Bowel Disease
* Inability to schedule the colonoscopy within 60 days of the initial stool sample
* Colonic pathology that in the opinion of the endoscopist could interfere with the accuracy of the colonoscopy. Examples include: colonic stricture, poor preparation, obstructing tumor.
* ASA class 4 or greater
* Vulnerable subjects. Students, nursing home residents, institutionalized patients, and those with psychological or physical incapacity.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at average risk of developing colorectal cancer, scheduled for colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Performance of Metabiomics Colon Polyp and Colorectal Cancer Assay | 1 year
  Microbiome based predictions from at least 100 blinded samples will be compared with colonoscopy and pathology results to quantify the sensitivity, specificity and accuracy (reported as %) of the Metabiomics Colon Polyp and Colorectal Cancer Assay for colon polyps. The limited sample size is anticipated to be insufficient to quantify sensitivity to colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hardi, M.D., Principal Investigator — Metropolitan Gastroenterology Group; Louis Korman, M.D., Principal Investigator — Metropolitan Gastroenterology Group
Locations (2):
- United States (2):
  - DC Endoscopy Center, Washington D.C., District of Columbia
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland

REFERENCES:
- See also: Click here for more information about the sponsor of this study, Metabiomics. — http://metabiomics.com/